CLINICAL TRIAL: NCT06292624
Title: Effectiveness of Intermittent Vacuum Therapy Combined with Aerobic Exercise in Improving Lower Limb Oxygenation and Circulation in Individuals with Diabetes Mellitus
Brief Title: Effectiveness of Intermittent Vacuum Therapy Combined with Aerobic Exercise in Individuals with Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Yan Chai Hospital Social Services (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20230417002
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm, receiving IVT combined with cycling exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intermittent vacuum therapy + Cycling exercise (Experimental): Participants received 12 IVT sessions of 30 minutes combined with 20 minutes of cycling exercise during the 6-week period.
  Interventions: Device: Intermittent vacuum therapy (Weyergans High Care® Medial, Germany); Behavioral: Cycling exercise

INTERVENTIONS:
Device: Intermittent vacuum therapy (Weyergans High Care® Medial, Germany) — The participants' lower limb will be placed in the vacuum chamber and sealed with a cuff. The maximum negative pressure applied in the experimental group would be -40mmHg (negative pressure/ambient pressure phase: 9s / 7s). The parameters are selected based on the manufacturer's recommendations.
Behavioral: Cycling exercise — The participant will perform 20 minutes of cycling exercise. Aiming at reaching a moderate exercise intensity (50% - 70%) of maximal heart rate on a gym bike.

SUMMARY:
Consequences of the compromised vascular system in diabetes mellitus (DM) are among the most devastating complications. Reduction in blood flow and oxygen uptake of skeletal muscle leads to muscle fatigue and impaired skeletal muscle post-exercise adaptation. Recent studies showed that intermittent vacuum therapy (IVT) augments the blood flow of the foot in people with DM. This pilot study investigates the effects of combined IVT and aerobic exercise in improving lower limb muscle oxygenation and distal circulation in individuals with DM. Positive results of the study shed light on strategy that enhances the effectiveness of aerobic exercise in people with DM.

DETAILED DESCRIPTION:
This study addresses the significant global health issue of Diabetes Mellitus (DM), a chronic condition characterized by the body's inability to properly use and store glucose. With an estimated 422 million adults affected worldwide in 2014, projected to increase to 629 million by 2045, DM poses a substantial public health challenge. Specifically, in Hong Kong, the prevalence was around 8.4% in 2014, and by 2021, DM had become the tenth leading cause of death. One of the most devastating complications of DM is the damage to the vascular system.

Recent developments in treatment options include Intermittent Vacuum Therapy (IVT), a technique initially developed for astronauts to mitigate orthostatic complications. IVT involves the application of alternating negative and ambient pressures to the lower extremities, which has been shown to enhance blood flow by promoting rhythmic vasodilation and compression. This method has successfully increased foot perfusion in both healthy volunteers and patients with Peripheral Artery Disease (PAD), highlighting its potential benefits in improving circulation without direct contact with the patient's limb, thereby minimizing the risk of cross-infection.

The study also explores the role of aerobic exercise in improving insulin sensitivity, blood sugar control, and reducing DM-related complications. However, DM patients often face challenges such as muscle fatigue during exercise due to impaired glucose uptake, mitochondrial dysfunction, microvascular damage, and atherosclerosis, which limit blood supply to skeletal muscles, affecting exercise capacity.

Given the positive effects of IVT on distal circulation in PAD patients but its unexplored benefits in DM patients when combined with aerobic exercise, the study hypothesizes that IVT could enhance distal circulation, oxygen uptake, and nutrient delivery to the skeletal muscle of the lower limbs. This could, in turn, amplify the benefits of aerobic training on skeletal muscle in DM patients.

The study's objectives are twofold:

To evaluate the feasibility, safety, and patient acceptance of combining IVT with an exercise program in DM rehabilitation.

To examine the effectiveness of this combined approach on lower-limb perfusion, muscle physiology, and locomotion functions in DM patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 55 and 80 years old,
* being diagnosed with Type 2 DM,
* being able to give informed consent to participate in the study.
* able to walk without assistance

Exclusion Criteria:

* have a conditions that contraindications to IVT: pregnancy, abdominal wall hernia, recent (<8 weeks) trauma of the lower limbs,
* have an open wound on the lower extremity or with lower extremity infection,
* have any orthopaedic or medical conditions that could hinder the assessment and training.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Muscle oxygenation | baseline
  Two wireless NIRS (Near-infrared Spectroscopy) sensors (Portamon, Artinis Medical Systems,The Netherlands) will be placed on participants' dorsal feet and quadriceps on their dominant leg. The signal will be collected continuously for 10 minutes during cycling.
Muscle oxygenation | post-treatment (6weeks)
  Two wireless NIRS sensors (Portamon, Artinis Medical Systems,The Netherlands) will be placed on participants' dorsal feet and quadriceps on their dominant leg. The signal will be collected continuously for 10 minutes during cycling.

SECONDARY OUTCOMES:
Surface Electromyography | baseline
  Muscle fatigue of the quadriceps and calf muscles during cycling exercise will be quantified by the median frequency and mean power frequency extracted from surface electromyography signal.
Surface Electromyography | post-treatment (6weeks)
  Muscle fatigue of the quadriceps and calf muscles during cycling exercise will be quantified by the median frequency and mean power frequency extracted from surface electromyography signal.
Foot Sensation | baseline
  The monofilament test, which involves pointing a nylon filament over various areas of the foot to test for the ability to detect light touch, will be used to assess the foot sensory. It is considered a reliable method to detect the presence of peripheral neuropathy.
Foot Sensation | post-treatment (6weeks)
  The monofilament test, which involves pointing a nylon filament over various areas of the foot to test for the ability to detect light touch, will be used to assess the foot sensory. It is considered a reliable method to detect the presence of peripheral neuropathy.
Functional muscle strength | baseline
  The functional muscle strength will be assessed by the Five-Time Sit-to-Stand Test.The functional muscle strength will be assessed by the Five-Time Sit-to-Stand Test. Assessing the completion time of 5 sit-to-stand movement.
Functional muscle strength | post-treatment (6weeks)
  The functional muscle strength will be assessed by the Five-Time Sit-to-Stand Test. Assessing the completion time of 5 sit-to-stand movement.
Functional mobility | baseline
  Functional mobility will be assessed by the Timed Up and Go Test
Functional mobility | post-treatment (6weeks)
  Functional mobility will be assessed by the Timed Up and Go Test

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to other researchers